CLINICAL TRIAL: NCT01757210
Title: A Study to Evaluate the Safety and Efficacy of Aprepitant (MK0869) for Chemotherapy-Induced Nausea and Vomiting in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: West Virginia University Healthcare (Other)
Responsible Party: Principal Investigator, Lisa Biondo, Pharm.D., BCPS, West Virginia University Healthcare
Other Study IDs: 24267
Record Dates: First submitted 2012-09-27; First posted 2012-12-28 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
Keywords: Aprepitant; Pediatrics; Chemotherapy-induced nausea/vomiting; Survey
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aprepitant was approved in 2003. The drug works to lessen the amount of nausea and vomiting that cancer patients experience after treatment. Aprepitant has been well-studied in adults, but not in children. Data from adult studies has shown aprepitant to be safe. It has also been shown to be effective in lessening the amount of nausea and vomiting that adult patients experience. Because aprepitant has been shown to be safe and effective, the investigators have been using it in pediatric patients at this hospital as standard of care. The investigators will be surveying patients already receiving aprepitant for prevention of chemotherapy-induced nausea and vomiting to determine the amount of nausea and vomiting they experience. The investigators will also be surveying these patients to determine what their appetite is like and if they experience any disruptions in activities of daily living. The investigators are also going to be assessing any side effects these patients experience from receiving aprepitant.

DETAILED DESCRIPTION:
This will be a prospective, observational study conducted at WVU Children´s Hospital. The study will be conducted over a one-year period until data from 20-40 patient encounters is obtained. There will be no randomization and no control group. Information will be collected from all patients who meet the study´s inclusion criteria. Patients will be given a survey to complete at baseline, on all days of chemotherapy, and for five days after the conclusion of chemotherapy using the BARF Scale and a 4-point Likert scale. The information collected from the survey will include the incidence and severity of nausea and emesis, evaluation of appetite, activities of daily living, and rescue medications used for acute CINV. The specific chemotherapy regimen that each patient receives will be recorded. Any data identifying the patient will be de-identified after all pertinent data is collected. Descriptive statistics will be used to analyze data.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between the ages of 1-17 years
2. Patient has a confirmed malignancy
3. Patient is receiving highly or moderately emetogenic chemotherapy
4. Receiving aprepitant as part of an anti-emetic regimen
5. Patient's legally-authorized representative understands and voluntarily signs the written informed consent prior to any study-specific procedures. A copy of the signed informed consent form will be retained by the treating institution.
6. Patient ≥7 years of age understands and voluntarily signs the written informed assent form prior to any study specific procedures. A copy of the signed informed assent form will be retained by the treating institution.

Exclusion criteria:

1. Pregnant or breast feeding
2. Concomitant use of pimozide, terfenadine, astemizole, or cisapride
3. Child-Pugh score > 9
4. Receiving IV fosaprepitant

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will include pediatric patients with an active malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of episodes of nausea and vomiting | Five days after end of chemotherapy
  The primary outcome measure is assessing the incidence of chemotherapy-induced nausea and vomiting in pediatric patients receiving highly or moderately emetogenic chemotherapy and a prophylactic regimen that includes aprepitant. The incidence of chemotherapy-induced nausea and vomiting will be evaluated using the BARF Scale and a 4-point Likert scale on all days of chemotherapy and for five days following the conclusion of chemotherapy compared to baseline

SECONDARY OUTCOMES:
Appetite score on a 4-point Likert scale | Five days after the end of chemotherapy
  Patients will be assessed for changes in appetite using a 4-point Likert scale at baseline, on all days of chemotherapy, and for the five days following the conclusion of chemotherapy
Activities of daily living score on a 4-point Likert scale | Five days after the end of chemotherapy
  Patients will be assessed for changes in activities of daily living using a 4-point Likert scale at baseline, on all days of chemotherapy, and for five days following the conclusion of chemotherapy
Number of medications used for breakthrough nausea and vomiting | Five days after the end of chemotherapy
  The usage of all breakthrough medications for chemotherapy-induced nausea and vomiting while in the hospital will be recorded.
Participants with Adverse Events as a Measure of Safety and Tolerability | Five days after the end of chemotherapy
  Incidence of adverse events that can be definitely or probably related to aprepitant using the Naranjo Adverse Event Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Biondo, Pharm.D., Principal Investigator — WVU Healthcare
Locations (1):
- WVU Healthcare, Morgantown, West Virginia, United States

REFERENCES:
- [Background] Smith AR, Repka TL, Weigel BJ. Aprepitant for the control of chemotherapy induced nausea and vomiting in adolescents. Pediatr Blood Cancer. 2005 Nov;45(6):857-60. doi: 10.1002/pbc.20378. PMID 15849684
- [Result] Choi MR, Jiles C, Seibel NL. Aprepitant use in children, adolescents, and young adults for the control of chemotherapy-induced nausea and vomiting (CINV). J Pediatr Hematol Oncol. 2010 Oct;32(7):e268-71. doi: 10.1097/MPH.0b013e3181e5e1af. PMID 20736848
- [Result] Gore L, Chawla S, Petrilli A, Hemenway M, Schissel D, Chua V, Carides AD, Taylor A, Devandry S, Valentine J, Evans JK, Oxenius B; Adolescent Aprepitant in Cancer Study Group. Aprepitant in adolescent patients for prevention of chemotherapy-induced nausea and vomiting: a randomized, double-blind, placebo-controlled study of efficacy and tolerability. Pediatr Blood Cancer. 2009 Feb;52(2):242-7. doi: 10.1002/pbc.21811. PMID 18985740